CLINICAL TRIAL: NCT00055055
Title: Pathogenic Studies In Families With Twins Or Siblings Discordant For Systemic Rheumatic Disorders
Brief Title: Study of Families With Twins or Siblings Discordant for Rheumatic Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030099; 03-E-0099
Record Dates: First submitted 2003-02-15; First posted 2003-02-17 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-05-20

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus; Idiopathic Inflammatory Myopathies
Keywords: Autoimmunity Pathogenesis; Microarray Analyses; Microchimerism; Natural History
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Myositis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Healthy Volunteers: A healthy individual who has not used any NSAIDS, with no infectious disease, or severe trauma within 8 weeks of enrollment, doesn't have a first degree relatives with RA, SLE, SSc or IIM
- Parent of Proband: Biological mother or father of the proband who is willing to enroll in the study
- Primary Unaffected Dizygous Twin: Dizygotic twin pair of the proband who does not meet criteria for one of the rheumatic diseases
- Primary Unaffected Monozygous Twin: Monozygotic twin pair of the proband who does not meet criteria for one of the rheumatic diseases
- Primary Unaffected Non-twin Sibling: Sibling of the same biological parents, same gender, within 5 years of age of the proband who does not meet criteria for one of the rheumatic diseases
- Proband: Proband should have documented evidence that he/she meets criteria for adult and juvenile forms of systemic rheumatic disorders

SUMMARY:
This study will examine families in which one sibling of a sibling pair, or twin pair, has developed a systemic rheumatic disease and one has not, to see if and how the two differ in the following:

* Blood cell metabolism;
* Types of cells in the blood;
* Environmental exposures or genetic factors that might explain why one developed disease and the other did not.

Families in which one sibling has developed a systemic rheumatic disease, rheumatoid arthritis, systemic lupus erythematosus, scleroderma, dermatomyositis, or myositis, and the other has not, are eligible for this study. The siblings may or may not be twins, but must be of the same gender and be within a 5-year age difference. Biological parents, or, in some cases, children, will also be included in the study. Normal, healthy volunteers will serve as control subjects.

Participants will undergo some or all of the following tests and procedures:

* Medical history and physical examination. Participants will also be asked permission to obtain medical records for review.
* Questionnaires about environmental exposures at work, at home, and elsewhere. Probands (participants with rheumatic disease) and their healthy siblings will also answer questions about infections, vaccinations, medications or dietary supplements, sun exposure, and stressful events during the year before disease diagnosis in the affected sibling.
* Blood and urine collection for the following tests:
* Routine blood chemistries and other studies to rule out certain diseases or medical problems;
* Evidence of past toxic exposures and certain infections;
* Presence of cells from the mother in the child s blood and vice versa. (Recent studies suggest that during pregnancy or delivery, cells from the mother and baby may be exchanged and circulate in the body for many years, possibly causing problems);
* In twin or sibling pairs, presence of certain genes that may be more common in patients with systematic rheumatic diseases as compared with their unaffected siblings and normal volunteers;
* In identical twins, comparison of their blood cell metabolism to see if and how the metabolism differs in people with rheumatic disease.

Participants may be asked for permission to have some of their blood and urine samples stored and to obtain previously collected blood or tissue biopsy specimens that are no longer needed for clinical care, for research purposes. They may also be asked to give additional blood or urine samples.

Participants will be followed every year for 5 years (either in person or by questionnaire) to evaluate any changes in their condition. The final 5-year evaluation will repeat some of the questionnaires and procedures described above.

DETAILED DESCRIPTION:
Most autoimmune diseases are thought to develop as a result of chronic immune activation and dysregulation after selected environmental exposures in genetically susceptible individuals. Current evidence suggests that the adult and juvenile forms of systemic rheumatic disorders -- defined here as rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), systemic sclerosis (SSc), and idiopathic inflammatory myopathies (IIM) -- share many common clinical manifestations, immune responses, genetic, hormonal and environmental risk factors, and possible pathogeneses. Conversely, other studies imply that each rheumatic disease, as currently defined, may be composed of more homogeneous subgroups, known as elemental disorders, with different pathogeneses. This protocol will explore pathogenic mechanisms for systemic rheumatic disorders and possible elemental disorders through the evaluation of families with monozygotic or dizygotic twins or other siblings discordant for systemic rheumatic disorders (twin-sib pairs). Parents and healthy volunteers will also be evaluated as needed for the experimental designs of each portion of the protocol. A clinical evaluation, using standardized physician and patient clinical and environmental exposure questionnaires, and specimen collections from 400 twin-sib pairs discordant for systemic rheumatic disorders will be performed to confirm diagnoses, document medical histories and assess possible risk factors implicated in the development of autoimmunity. This study will evaluate children, who will make up 25-50% of the twin-sib pairs, and adults in similar ways to attempt to understand possible similarities and differences in pathogeneses of systemic rheumatic disorders based upon age of onset. Hypothesis-testing studies will assess differences in peripheral blood cell gene activation/suppression, levels and types of microchimerism between affected and unaffected individuals, selected genetic risk factors for these disorders and occupational and hormonal exposures hypothesized to be potential risk factors for these diseases. Exploratory studies will be conducted to begin to assess other environmental risk factors for systemic rheumatic disorders and to better understand associations among phenotypes and genotypes. Biologic specimens -- including blood, urine, and other clinical specimens or biopsies no longer necessary for clinical care -- will be collected for directed biomarker assays and the development of repositories for future research.

ELIGIBILITY:
* INCLUSION CRITERIA:

The minimum inclusion criteria needed for enrollment are a twin pair or sibling pair, as defined by an eligible proband and his/her eligible twin or sibling, willing and able to give informed consent, to enroll in the study, to complete the questionnaires and to donate blood and urine samples (in case of children, parent/legal guardian must also be willing and able to provide informed consent).

Proband inclusion criteria:

- Children (< 18 years of age) or adults (18 or more years of age) require a diagnosis of a systemic rheumatic disorder (by American College of Rheumatology (ACR) or other criteria for the adult or juvenile forms of RA, SLE, SSc, or IIM (per (92;93)). Regarding the childhood-onset diseases: JRA will be defined by age of onset <17 years of age; for other diseases age of onset will be < 18 years. Probands will be diagnosed within 5 years of enrollment in the study, with at least one twin or other sibling of the same gender within 5 years of age and without a recognized systemic rheumatic disorder or other autoimmune disease available for study.

Twin-sibling inclusion criteria:

-Children or adults who are twins or other siblings of a proband sharing the same biological parents, but without a recognized systemic rheumatic or autoimmune disorder, of the same gender and within 5 years of age of the proband. If monozygotic twins are enrolled from a family, another unaffected non-twin sibling sharing the same biological parents will be enrolled for each proband if available to allow for log-linear genetic analyses. All probands and unaffected siblings need to be at least one year of age at the time of autoimmune disease diagnosis. In the case of triplets or greater multiples, all such siblings are eligible for enrollment.

Parent inclusion criteria:

-Individuals who are the genetic father and mother of the proband and twin-sib. Both parents will be enrolled whenever possible.

Healthy volunteer inclusion criteria:

Healthy controls, recruited in part via the NIH Healthy Volunteers program, and as reasonably as possible, matched to a subset of probands based on age (within 5 years), gender, and race (when feasible). Healthy volunteers should be in good health, without

a recognized systemic rheumatic disorder or other autoimmune disease, and should not be taking antiinflammatory medicines, including nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids.

For all subjects: ability of the subject or parents/legal guardians to provide informed consent to all aspects of the study after full protocol information is provided.

Should a participant enroll at a time when his/her twin/sibling is willing and able to give informed consent, but his/her twin/sibling never enrolls (eg. Due to no longer being willing or able to give informed consent), the enrolled participant will remain in the study and his/her data will be used in the analyses not pertinent to his/her twin/sibling. Data analysis will also occur in this manner should the enrolled participant s sibling enroll, but never send in blood samples and/or questionnaires.

EXCLUSION CRITERIA:

Exclusion criteria for all protocol subjects:

1. severe trauma or vaccinations within 8 weeks of enrollment;
2. Still s disease/systemic-onset or pauciarticular JRA;
3. medical illness that in the judgment of the investigators does not allow safe blood draws or other clinical evaluations needed for study participation;
4. cognitive impairment;
5. inability to give informed assent or consent.

Exclusion criteria for twin-sibs:

Not sharing the same biological parents (being half-brothers or half-sisters). Known criteria for systemic rheumatic disease or autoimmune disease (for example: RA/JRA, SLE/JSLE, SSc/JSSc, IIM/JIIM, Type 1 diabetes, Psoriasis, Still s disease/systemic-onset or pauciarticular JRA, Celiac sprue, Autoimmune thyroid disease, Idiopathic Thrombocytopenia Purpura, Multiple sclerosis, Myasthenia gravis, Systemic vasculitis or Vitiligo).

Exclusion criteria for healthy volunteers:

Recognized systemic rheumatic disorder or other autoimmune disease, history of cancer or taking anti-inflammatory medicines, including nonsteroidal anti-inflammatory drugs (NSAIDs) or corticosteroids, severe trauma or vaccinations within 8 weeks.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1- Proband who have documented evidence that he/she meets criteria for adult and juvenile forms of systemic rheumatic disorders defined here as rheumatoid arthritis (RA), systemic lupus 2- Twin pair of the proband who does not meet criteria for one of the rheumatic diseases and is willing to give consent and enroll in the study 3- Sibling of the same biological parents, same gender, within 5 years of age of the proband who does not meet criteria for one of the rheumatic diseases and is willing to give consent and enroll in the study 4- Biological mother or father of the proband who is willing to enroll in the study 5- A healthy individual who has not used any anti-inflammatory medications, has not had an infectious disease(persistent or chronic infection, history of M. tuberculosis, HIV or active infection), or experienced severe trauma within 8 weeks of enrollment, doesn't have a first degree relatives with RA, SLE, SSc or IIM and is willing to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 1056 (Actual)
Dates: Start 2003-04-21 (Actual)

PRIMARY OUTCOMES:
Physician Global Assesment Questionnaire | At enrollment and each study
  Evaluate core set disease activity, damage and quality of life measures in adult and juvenile myositis patients

CONTACTS AND LOCATIONS:
Overall Officials: Lisa G Rider, M.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NIEHS Clinical Research Unit (CRU), Research Triangle Park, North Carolina
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan for IPD availability, we are still deciding

REFERENCES:
- [Background] Gan L, O'Hanlon TP, Gordon AS, Rider LG, Miller FW, Burbelo PD. Twins discordant for myositis and systemic lupus erythematosus show markedly enriched autoantibodies in the affected twin supporting environmental influences in pathogenesis. BMC Musculoskelet Disord. 2014 Mar 6;15:67. doi: 10.1186/1471-2474-15-67. PMID 24602337
- [Background] O'Hanlon TP, Rider LG, Gan L, Fannin R, Paules RS, Umbach DM, Weinberg CR, Shah RR, Mav D, Gourley MF, Miller FW. Gene expression profiles from discordant monozygotic twins suggest that molecular pathways are shared among multiple systemic autoimmune diseases. Arthritis Res Ther. 2011 Apr 26;13(2):R69. doi: 10.1186/ar3330. PMID 21521520
- [Background] Javierre BM, Fernandez AF, Richter J, Al-Shahrour F, Martin-Subero JI, Rodriguez-Ubreva J, Berdasco M, Fraga MF, O'Hanlon TP, Rider LG, Jacinto FV, Lopez-Longo FJ, Dopazo J, Forn M, Peinado MA, Carreno L, Sawalha AH, Harley JB, Siebert R, Esteller M, Miller FW, Ballestar E. Changes in the pattern of DNA methylation associate with twin discordance in systemic lupus erythematosus. Genome Res. 2010 Feb;20(2):170-9. doi: 10.1101/gr.100289.109. Epub 2009 Dec 22. PMID 20028698
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2003-E-0099.html